CLINICAL TRIAL: NCT04140604
Title: A Three-arm, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety of Lactobacillus Salivarius AP-32 and Bifidobacterium Animalis Subsp. Lactis CP-9 Used Individually in Healthy Infants
Brief Title: Safety Evaluation of Lactobacillus Salivarius AP-32 and Bifidobacterium Animalis Subsp. Lactis CP-9 in Healthy Infants.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hsieh-Hsun Ho (Industry)
Responsible Party: Sponsor-Investigator, Hsieh-Hsun Ho, R.D. Senior Manager, Glac Biotech Co., Ltd
Organization: Glac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GLA-001
Record Dates: First submitted 2019-10-22; First posted 2019-10-28 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Safety Issues
Keywords: Probiotic; Lactobacillus salivarius AP-32; Bifidobacterium animalis subsp. lactis CP-9; Safety; Healthy infant

STUDY DESIGN:
Intervention Model Description: Active:
  1. Lactobacillus salivarius AP-32.
  2. Bifidobacterium animalis subsp. lactis CP-9. supplied as 0.5 g capsules.
  Placebo:
  The placebo capsules are identical to the Lactobacillus salivarius AP-32 and Bifidobacterium animalis subsp. lactis CP-9 capsules except for the probiotics.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study so neither investigator and site staff, nor the subject know which treatment has been assigned.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lactobacillus salivarius AP-32 (Experimental): A 0.5 g light-yellow capsule containing freeze-dried powder of 2.5 billion CFU of Lactobacillus salivarius AP-32 and maltodextrin.
  Interventions: Other: Lactobacillus salivarius AP-32
- Bifidobacterium animalis subsp. lactis CP-9 (Experimental): A 0.5 g light-yellow capsule containing freeze-dried powder of 2.5 billion CFU of Bifidobacterium animalis subsp. lactis CP-9 and maltodextrin.
  Interventions: Other: Bifidobacterium animalis subsp. lactis CP-9
- Placebo (Placebo Comparator): The placebo composition and appearance are the same as probiotic capsules, but does not contain live bacteria.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Lactobacillus salivarius AP-32 — Infants will be given the content of one capsule (mixed in infant formula or breast milk) twice daily (morning and evening) for 15 weeks.
  Arms: Lactobacillus salivarius AP-32
Other: Bifidobacterium animalis subsp. lactis CP-9 — Infants will be given the content of one capsule (mixed in infant formula or breast milk) twice daily (morning and evening) for 15 weeks.
  Arms: Bifidobacterium animalis subsp. lactis CP-9
Other: Placebo — Infants will be given the content of one capsule (mixed in infant formula or breast milk) twice daily (morning and evening) for 15 weeks.
  Arms: Placebo

SUMMARY:
This is a three-arm, double-blind, placebo-controlled study to investigate the safety of Lactobacillus salivarius AP-32 and Bifidobacterium animalis subsp. lactis CP-9 used individually in healthy infants.

Infants will be given the content of one capsule (mixed in infant formula or breast milk) twice daily (morning and evening) for 15 weeks.

DETAILED DESCRIPTION:
This is a three-arm, double-blind, placebo-controlled study to investigate the safety of Lactobacillus salivarius AP-32 and Bifidobacterium animalis subsp. lactis CP-9 used individually in healthy infants.

Infants will be given the content of one capsule (mixed in infant formula or breast milk) twice daily (morning and evening) for 15 weeks. Follow-up visits will take place at study days 14±3, 42±3, 70±4 and 105±4.

Caregivers will keep a diary of the volume of formula intake/minutes of breastfeeding, stool frequency and consistency (hard, formed, soft/paste or loose/watery), symptoms of digestive tolerance (regurgitation and flatulence), sleeping time, crying/fussing time and episodes for 3 days before each visit. At each visit, the research team will review the diary and conduct physical examination, including anthropometric measurements (weight, recumbent length, and head circumference).

Fecal samples will be collected prior to the first administration of the assigned study product and at the end of study for microbiota analysis.

Adverse events (AEs) will be assessed based on inquires to the caregivers. AEs will be classified as related or unrelated based on a relationship to study product intake according to the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Having informed consent of the parent or legal guardian.
* Healthy male and female infants between 7 days and 2 months (60 ± 2 days) of age at the time of study initiation.
* Full term ( ≧ 36 weeks gestation at birth).
* Birth weight ≧ 2500 g.
* Able and willing to comply with all study requirements.

Exclusion Criteria:

* Failure to thrive (weight gain < 100 grams/week average from birth to the last recorded weight).
* Major acute or chronic illness (e.g. significant cardiac, respiratory, hematological, gastrointestinal or other systemic diseases, major developmental or genetic abnormality).
* Use of substances that alter gut microbiota (antibiotics, prebiotics, probiotics or gastric acid inhibitors) within 2 weeks prior to the study initiation.
* For breastfed infants, use of antibiotics, prebiotics and probiotics by the mothers.
* Cow's milk protein allergy.
* Feeding difficulties.
* History of any allergies to maltodextrin.
* Participation in another clinical trial.
* Any other clinically significant medical, psychiatric and/or social reason as determined by the investigator.

Ages: 7 Days to 60 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Mean weight gain. | 15 weeks.
  The change value from baseline at the end of the treatment.

SECONDARY OUTCOMES:
Occurrence of adverse events (AEs). | 15 weeks.
  The occurrence of adverse events (AEs) during the period of probiotic or placebo intervention.
Anthropometric measurements of recumbent length. | 15 weeks.
  The change value from baseline at the end of the treatment.
Anthropometric measurements of head circumference. | 15 weeks.
  The change value from baseline at the end of the treatment.
Incidence of regurgitation. | 15 weeks.
  Caregivers will be instructed by the investigator or the designated study center personnel to record the regurgitation for three days within the week before each study visit. At each study visit, the investigator or the designated study center personnel will review the diary and record the times of regurgitation.
Incidence of flatulence. | 15 weeks.
  Caregivers will be instructed by the investigator or the designated study center personnel to record the flatulence for three days within the week before each study visit. At each study visit, the investigator or the designated study center personnel will review the diary and record the times of flatulence.
Incidence of infectious diseases. | 15 weeks.
  Observing the incidence of infectious diseases during the period of probiotic or placebo intervention.
Incidence of allergic diseases. | 15 weeks.
  Observing the incidence of allergic diseases during the period of probiotic or placebo intervention.
Crying and/or fussing time (hours/day) and episodes. | 15 weeks.
  Observing the crying and/or fussing time (hours/day) and episodes during the period of probiotic or placebo intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hsieh-Hsun Ho, Ph.D, Principal Investigator — Glac Biotech Co., Ltd
Locations (1):
- Glac Biotech Co., Ltd, Tainan, Taiwan